CLINICAL TRIAL: NCT05832814
Title: The Effect of Music Therapy in Pulmonary Rehabilitation of COPD Patients Aged 40-75
Brief Title: Music Therapy for COPD Rehabilitation
Acronym: COPDMELODY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Ting YANG, Principal Investigator, Clinical Professor, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-HX-16
Record Dates: First submitted 2022-07-31; First posted 2023-04-27 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; music therapy; pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Integrated training (Experimental): Rhythm-guided walking exercise coordinated with singing training as training activity in pulmonary rehabilitation: 12 weeks, three times a week for 1 hour, leading to a total of 36 sessions
  Interventions: Behavioral: Integrated training
- Rhythm-guided exercise training (Experimental): Rhythm-guided walking exercise as training activity in pulmonary rehabilitation: 12 weeks, three times a week for 1/2 hour, leading to a total of 36 sessions
  Interventions: Behavioral: Rhythm-guided exercise training
- Usual care (No Intervention): The usual care is the comparator in the trial, consisting of standard medical treatment and educational sessions including physical training, smoking cessation and vaccination. And after the trial, the patients in this group will also be offered standard pulmonary rehabilitation according to the national guideline.

INTERVENTIONS:
Behavioral: Integrated training — For rhythm-guided walking exercise, the home exercise intensity, that is, the walking speed can be prescribed based on the incremental shuttle walking(ISWT) result. A rhythm matching with the walking speed can be calculated. Then patients will be provided a group of melodies identified by the calculated rhythm, which are also popular with the elder. During exercise, the patients are required to walking on a fixed speed identical with the rhythm. For singing training, patients follow the audios and videos to take training at home, which are recorded by singing teachers and physiotherapists prior to the trial. Each session includes technical instructions in order to achieve better respiratory control during singing.
  Arms: Integrated training
Behavioral: Rhythm-guided exercise training — For rhythm-guided walking exercise, the home exercise intensity, that is, the walking speed can be prescribed based on the incremental shuttle walking test(ISWT) result. A rhythm matching with the walking speed can be calculated. Then patients will be provided a group of melodies identified by the calculated rhythm, which are also popular with the elder. During exercise, the patients are required to walking on a fixed speed identical with the rhythm.
  Arms: Rhythm-guided exercise training

SUMMARY:
Chronic obstructive pulmonary disease(COPD) patients could benefit from pulmonary rehabilitation(PR) in better managing of the disease and its symptoms and in avoiding future relapses and hospitalizations. However, due to a large number of drop outs from PR, lack of professionals, and the COVID-19 epidemic, the PR has been underutilized, leading to a need for investigation of updated forms. Music therapy, such as rhythm-guided endurance training, singing training, listening to melody, may be one such potential relevant and motivating rehabilitation activity. The study aims to investigate the effects of home-based PR program with a rhythm-guided endurance walking exercise and singing training on both physiological and psychological aspects. Effects will be investigated in a randomized controlled trial (RCT) with 12-week intervention period.

DETAILED DESCRIPTION:
Physiology and psychology of COPD

COPD is a syndrome with a progressive pulmonary obstruction leading to increasingly impaired lung function due to chronic inflammation in the respiratory passages and pulmonary tissue. Living with COPD everyday life is a struggle and often marked with reduced physical activity, again leading to progression of disease, by which a vicious circle develops. Declining physical performance is associated with ventilation restriction, insufficient oxygen diffusion, respiratory muscle and peripheral skeletal muscle dysfunction, ventricular dysfunction and so on.

On a psychological level COPD patients tend to suffer from comorbidities such as increased stress and anxiety levels e.g. due to dyspnea and dysfunction. In conclusion, COPD often leads to a severe condition that both physically and psychologically can be very difficult to manage and cope with.

COPD and rehabilitation

Pulmonary rehabilitation (PR) is multidisciplinary and comprehensive intervention that may improve the interrelated physical and psychological consequences of the disease. It is designed to optimize functional status, reduce symptoms, improve health-related quality of life, reduce anxiety and depression, reduce exacerbations and mortality. However, in spite of documented efficacy and strong recommendations, PR is largely underutilized because most programs have been carried out on an inpatient or outpatient basis, relying on high cost, adequate doctors or therapists and regular visits to hospital. Another problem is the long-term maintenance of benefits once the hospital-based PR program has been completed, since gains achieved diminish progressively if training is abandoned. For these reasons, home-based PR has been proposed as an alternative to outpatient rehabilitation.

Just like the supervised training, a home-based PR program must include endurance exercise training, e.g. walking. Optimally, a program should also include respiratory muscle training.

Reviewing previous relevant researches, the current common home-based PR models have several limitations. The compliance is still pretty poor, both due to fear of dyspnea and fragility during training and tiring of inflexible exercise form. There is also a concern about ensurance of the exercise intensity during a home-based PR. Therefore it is of high importance to develop alternative rehabilitation activities that are motivating and are perceived helpful for the participants. This study aims to investigate music therapy(MT) as a new complementary therapy, since MT has the potential to facilitate exercise training and strengthen motivation of rehabilitation activity, with both physiological and psychological effects.

Music therapy and COPD rehabilitation

A number of international studies have investigated the effects of MT in relation to COPD patients. Music therapy targeting at COPD patients include offering music during exercise(distractive auditory stimulus therapy) and singing training. Compared with traditional aerobic exercise, rhythm-guided endurance training has the potential to help patients achieve a higher workload through decreasing or delaying the perception of exercise-induced dyspnea and fatigue. In terms of singing training, it could help patients learn how to control the respiratory function, including training and coordination of the related inspiratory and expiratory musculature. Moreover, from a psychology perspective, music in general seems to have an ability to promote motivations, and have a positive impact on well-being, anxiety and depression level.

Previous studies differ in methodology, and furthermore sample size and statistical power are not sufficient to conclude on significance and results. Most relevant researches are carried out in hospital or community-based face-to-face monitoring classes. No study has explored the integrated effects of music-facilitated exercise and singing training, although they might benefit COPD patients further through different physiological mechanisms compared with being applied separately. Therefore the present study is of high prevalence. Since it aims to develop alternative, motivating and personalized solutions to supplement standard PR, exploring whether singing training combined with melody-guided endurance exercise confers further benefits in exercise capacity and how music therapy influences patients' exercise performance, respiratory muscle strength, dyspnea, spirometry, quality of life and emotions.

ELIGIBILITY:
Inclusion Criteria:

Participants with a clinical diagnosis of COPD and meeting the following criteria are eligible:

1. Diagnosis of GOLD II-IV and without acute exacerbation within the last 4 weeks.
2. Motivated for participating in the project (and acceptance of randomization)
3. Sufficient mobility to attend PR

Exclusion Criteria:

1. Certain comorbidities (e.g. unstable coronary complications)
2. Severe cognitive disabilities (e.g. dementia)
3. Inability to cope with the program because of severe hearing or visual disorder.

No previous singing experience or musical competence is required.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
incremental shuttle walking test(ISWT) distance | 12 weeks
  incremental shuttle walking test distance

SECONDARY OUTCOMES:
Respiratory muscle strength | 12 weeks
  maximum inspiratory pressure(MIP), maximum expiratory pressure(MEP)
Spirometry | 12 weeks
  FEV1, FVC, FEV1/FVC, PEF, IC, RV, FRC, TLC
Short Physical Performance Battery(SPPB) | 12 weeks
  Test for health-related physical performance
modified British medical research council(mMRC) | 12 weeks
  It is a self-reported symptom questionnaire ranging from 0-4 score, higher scores mean a worse outcome.
COPD assessment test(CAT) | 12 weeks
  It is a self-reported quality of life questionnaire ranging from 0-10 score, higher scores mean a worse outcome.
St. George's Respiratory Questionnaire (SGRQ) | 12 weeks
  It is a self-reported symptom questionnaire ranging from 0-100 score, higher scores mean a worse outcome.
International Physical Activity Questionnaire Short Form (IPAQ-short) | 12 weeks
  It is a questionnaire evaluating participants' quantity of physical activity in a recent week.
Hospital Anxiety and Depression Scale(HADS) | 12 weeks
  It is a self-reported psychological status questionnaire ranging from 0-42 score, higher scores mean a worse outcome.
Compliance | 12 weeks
  Self-produced sheet with registration each time of each participant's attendance or absence (with or without cause). Registered continuously during intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Minghui Shi, MSc, Study Director — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Shi M, Yang L, Qumu S, Lei J, Huang K, He R, Niu H, Dong F, Wang S, He J, Yang T. Efficacy and safety of a music-therapy facilitated pulmonary telerehabilitation program in COPD patients: the COPDMELODY study protocol. Front Med (Lausanne). 2024 Mar 8;11:1361053. doi: 10.3389/fmed.2024.1361053. eCollection 2024. PMID 38523907